CLINICAL TRIAL: NCT04500288
Title: The Effect of Positional Therapy on Symptoms of Gastroesophageal Reflux Disease: A Prospective Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, RONNIE FASS, Ronnie Fass, MD, FACG, Director, Division of Gastroenterology and Hepatology, Head, Esophageal and Swallowing Center, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB20-00150
Record Dates: First submitted 2020-07-10; First posted 2020-08-05 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Gastro Esophageal Reflux
Keywords: Nocturnal Gastroesophageal Reflux Disease; Gastroesophageal Reflux Disease; LEFT Device; Sleep Hygiene
MeSH Terms: conditions — Gastroesophageal Reflux; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: This is a single center prospective Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEFT Device Arm (Experimental): Subjects in this arm will wear the LEFT device for 1 month
  Interventions: Device: LEFT Device

INTERVENTIONS:
Device: LEFT Device — LEFT device is a novel electronic wearable device that was developed as a sleep position therapy for patients who suffer from nighttime gastroesophageal reflux symptoms. It is simple, noninvasive and low-cost technology which has been developed by Side Sleep Technologies B.V. Singel, Amesterdam, The Netherland.
  Other Names: Epworth Sleepiness Scale; Sleep Quality Questionnaire; Berlin Questionnaire; Demographics Questionnaire; SF-36 Questionnaire; GERD symptoms checklist

SUMMARY:
Gastroesophageal reflux disease related symptoms are reported by 10-20% of the adult population and of those 50-75% report symptoms during sleep time. The prevalence of nocturnal GERD (nGERD) is estimated to be about 25% in general population. nGERD causes sleep fragmentation, difficulty falling asleep, daytime sleepiness, reduced work productivity and decreased quality of life. Additionally, nighttime gastroesophageal reflux has been associated with increased risk of GERD-related complications such as severe erosive esophagitis, peptic stricture, esophageal ulcer, Barrett's esophagus, and esophageal adenocarcinoma. Furthermore, nocturnal gastroesophageal reflux has been noted to be associated with atypical and extra-esophageal manifestations as well as sleep disturbances. Overall, patients with nocturnal gastroesophageal reflux are more likely to develop a more severe form of GERD. The mainstay of treatment of nighttime gastroesophageal reflux is a proton pump inhibitor (PPI). However, nighttime heartburn is the most common breakthrough symptom in patients with GERD, who failed PPI treatment. Other important therapies for nighttime GERD include, lifestyle modifications, such as elevating the head of the bed, avoiding eating at least three hours before bedtime, maintaining appropriate sleep hygiene and avoiding the right decubitus position. Elevating the upper torso by raising the head of the bed and avoiding the right-lateral decubitus position have been shown to improve nocturnal symptoms. Several studies have shown that sleeping in the left decubitus position decrease esophageal acid exposure by reducing 13-76% of the reflux episodes. Studies have shown that the right decubitus position increases the rate of transient lower esophageal sphincter relaxations (TLESRs) accompanied by acid reflux, as compared with the left recumbent position. Moreover, maintaining the left lateral recumbent position, reduced by 87% esophageal acid exposure and nocturnal symptoms.

LEFT is a novel electronic wearable device that was developed as a sleep position therapy for patients who suffer from nighttime gastroesophageal reflux symptoms. It is simple, noninvasive and low-cost technology which has been developed by Side Sleep Technologies B.V. Singel, Amesterdam, The Netherland.

This technology is designed to train patients to sleep on their left side by a gentle vibration signal once it detects that they are sleeping on their back or right side. Thus, this technique may reduce gastroesophageal reflux and thus provides relief of heartburn and regurgitation during sleep time. The purpose of this study is to determine the usefulness of positional therapy, using the LEFT device, as a nonmedical tool to control GERD-related nocturnal symptoms.

DETAILED DESCRIPTION:
Study Aims

1. The primary outcome of the study is to determine if positional therapy, using the LEFT device, is effective in improving nighttime GERD-related symptoms.
2. The secondary outcome of the study is to determine if positional therapy improves quality of sleep and health-related quality of life.

Methods:

Study Design This is a prospective, pilot study, that will be conducted at the Esophageal and Swallowing Center outpatient clinic at MetroHealth Medical Center. A total of 15 patients will be assessed for eligibility for the study. GERD patients will be recruited from the Esophageal and Swallowing Center outpatient clinic. Subjects with nighttime, GERD-related symptoms, at least three times a week will be recruited into the study. Nighttime symptoms are defined in this study as symptoms that awaken patients from sleep during the night. Subjects that meet inclusion and exclusion criteria will complete baseline pre-treatment validated questionnaires including, the Demographics Questionnaire, SF-36, GERD symptoms checklist, Berlin Questionnaire, Epworth Sleepiness Scale and Sleep quality questionnaire. Subsequently, patients will be trained on how to use the LEFT device. Prior to initiation of the study, the patients will undergo baseline symptoms assessment using the 7-day symptom record diary. Thereafter, patients will undergo positional therapy using the LEFT device for a period of one month. During the last week of the month, patients will undergo again the 7-day symptom record diary. On the last day of the month, patients will be asked to complete the following questionnaires, GERD symptoms checklist, Sleep quality questionnaire, and SF-36. The device well be returned together with the questionnaires by the patient.

Study population The study population will include patients with nocturnal GERD symptoms as previously defined, from our Esophageal and Swallowing Center outpatient clinic of MetroHealth Medical Center, main campus. Patients with at least three days of nighttime symptoms will be included in the study. Patients will be identified by clinical staff including attending physicians, GI fellows and Internal Medicine residents.

Patients seen in the Esophageal and Swallowing Center outpatient clinic will be identified if they appear to meet the study's inclusion and exclusion criteria. Patients will be contacted, followed, scheduled for appointments by the assigned research coordinator with input and advice as needed by the principal investigator.

Inclusion Criteria

1. Patients over the age of 18 who have proven GERD (with nighttime heartburn at least 3 days a week).
2. Agree to undergo sleep positioning therapy.
3. Able to read, understand, and complete study questionnaires.
4. Have mobile phones with an operating system (Android or iOS) that supports the LEFT device.

Exclusion Criteria

1. Patients who are under the age of 18.
2. Patients working night shifts.
3. Patients with significant comorbidity (cardiovascular, respiratory, renal, hematologic, endocrine, hepatic, gastrointestinal, neurological, or psychiatric).
4. Patients with history of major upper gastrointestinal surgery, active ulcer disease, existing diagnosis of esophageal motility disorder, systemic sclerosis, concomitant opiate use or diabetes mellitus.
5. Patients with obstructive sleep apnea

Study flow 15 Patients who meet the inclusion and exclusion criteria will be recruited into the study.

First visit - patients will receive baseline questionnaires including, Demographics Questionnaire, GERD symptoms checklist, Berlin Questionnaire, Epworth Sleepiness Scale, Sleep quality questionnaire and short form 36 (SF-36). In addition, patients will undergo 7- Day Symptom Record Diary.

Second visit - patients will be trained on how to use the LEFT device. Subsequently, patients will go through 10 days accommodation to the LEFT device. Thereafter, patients will use the LEFT device for one month. During the last week of the month, patients will undergo again the 7-day symptom record diary.

Third visit - On the last day of the month patients will fill again the GERD symptoms checklist, sleep quality questionnaire, SF-36, and return the LEFT device.

Demographics Questionnaire All subjects will complete a demographic questionnaire that evaluates age, education, employment, and annual household income. Data regarding alcohol and tobacco consumption will also be collected. Body Mass Index (BMI) will be calculated using an individual's height and weight.

GERD Symptoms checklist All subjects enrolled in the study will complete a validated GERD symptom questionnaire. This assesses the occurrence of heartburn, acid regurgitation, chest pain, trouble swallowing, and respiratory complaints. It will also assess esophageal abnormalities, surgical history, medication use and health-care utilization.

Berlin Questionnaire Berlin Questionnaire is used to assess risk factors for sleep apnea including the presence and frequency of snoring, wake-time sleepiness or fatigue, and obesity or hypertension. The questionnaire is composed of 15 questions divided among 3 different domains. Determination of the risk for obstructive sleep apnea is based on the responses to 3 different categories. In category 1, high risk is defined as persistent symptoms (more than 3 to 4 times per week) in 2 or more questions about snoring. In category 2, high risk is defined as persistent (more than 3 to 4 times a week) wake time sleepiness, drowsy driving, or both. In category 3, high risk is defined as history of high blood pressure or a BMI more than 30 kg/m2. To be considered a high risk for sleep apnea, a patient has to quality for at least 2 symptoms categories.

Epworth Sleepiness Scale (ESS) This is used for measure patient's subjective measure of a patient's sleepiness. The test is a list of eight situations in which patients rate their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. The total score is based on a scale of 0 to 24. The scale estimates whether patients are experiencing excessive sleepiness that possibly requires medical attention.

Sleep Quality Questionnaire (Sleep heart health study morning survey) This is validated questionnaire that was developed to determine sleep quality. The questionnaire assesses the previous night sleep. The questionnaire determines sleep quality by using 9 questions to assess and individual's perception of sleep quality and behaviors as they are related to quality of sleep. The questionnaire includes items such as "how many times did you awaken during night?" and "was your sleep restless or restful?" (rated on Linkert scales from 1 = restless to 5 = restful).

A subjective measure of overall sleep quality is calculated by using the responses from 5 items that are measured on a 5-point Linkert scale, summing them, and obtaining the average. In the following analysis, overall sleep quality is investigated in relation to other variables, and each item is also included separately in the analysis. Other variables assess the number of hours spent in bed, the number of hours slept, the number of awakenings, and the number of minutes that it took to fall asleep.

7- Day Symptom Record Diary

Patients will keep a daily record of the frequency and severity of each symptom they experienced for seven days. Symptoms such as daytime heartburn, nighttime heartburn, and acid regurgitation will be evaluated. The following scale will be used to determine severity of each symptom:

* Mild: Symptom easily tolerated and did not last long.
* Moderate: Symptom caused some discomfort but did not interfere with usual activities.
* Severe: Symptom caused much discomfort and interfered with usual activities. Disabling: Symptom unbearable and interfered considerably with usual activities.

SF-36 This is validated questionnaire that was developed to determine the overall health status. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 to 100. Lower score = more disability, higher scores = less disability.

Sections include, Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning and Mental health.

The LEFT device: LEFT is a novel reflux wearable device that is noninvasive and low-cost technology. The device was developed by Side Sleep Technologies B.V. Singel, Amesterdam, The Netherlands, as a sleep position therapy for patients who suffers from nighttime heartburn and other acid related symptoms. The technology is designed to train patients to sleep on their left side only during the night. The device tracks body position during sleep, then provides a gentle vibration signal once it detects that subjects are sleeping on their back or right side. This gentle vibration triggers the body to switch to the left side while asleep. During the adjustable period, the body may awaken from the gentle vibrations during the first 10 nights. While this may cause a minor sleep disruption as subjects adjust, it is important to continue to use the LEFT device in order to achieve the desired position effect.To ease the adjustment period, the LEFT device uses a specifically-designed pattern during the first 10 nights to progressively train the body to sleep on the left side.The device should be attached to the breastbone area by a disposable sticker that is replaced after each use. The LEFT device confirms its activation by vibrating 1 minute after being turned on and auto-start 20 minutes after being turned on, giving the patient time to fall asleep. The device also turns itself off automatically after 8 hours.

Data Collection:

Subjective symptom data will be collected from the questionnaires that patients will complete. The LEFT data will be downloaded from the device, collected and analyzed at MetroHealth Medical Center. Data will be stored in accordance with internal patient privacy rules as well as those of the IRB at our institution.

Statistical Analysis:

Unadjusted comparisons of continuous variables will be performed by appropriate parametric (t-test) and nonparametric (Mann-Whitney U test). Significant covariates such as age and gender will be adjusted for by employing multivariate regression models (SPSSv22). Data will be analyzed using prism and SPSS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18 who have proven GERD (with nighttime heartburn at least 3 days a week).
2. Agree to undergo sleep positioning therapy.
3. Able to read, understand, and complete study questionnaires.
4. Have mobile phones with an operating system (Android or iOS) that supports the LEFT device.

Exclusion Criteria:

1. Patients who are under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2024-05-21 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study is to determine if positional therapy, using the LEFT device, is effective in improving nighttime GERD-related symptoms as measured by GERD symptoms checklist (questionnaire, involves no specific units of measure). | 1 month
  Patients will undergo positional therapy using the LEFT device for a period of one month

SECONDARY OUTCOMES:
The secondary outcome of the study is to determine if positional therapy improves quality of sleep and health-related quality of life as measured by Epworth Sleepiness, Scale and Sleep quality, SF-36 and Berlin questionnaires. No units of measure. | 1 month
  Patients will undergo positional therapy using the LEFT device for a period of one month

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — Director, Division of Gastroenterology and Hepatology at Metrohealth MC; Abdulfatah Issak, MD, Principal Investigator — Gastroenterology Fellow at Metrohealth MC
Locations (1):
- Metrohealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Fass R, Quan SF, O'Connor GT, Ervin A, Iber C. Predictors of heartburn during sleep in a large prospective cohort study. Chest. 2005 May;127(5):1658-66. doi: 10.1378/chest.127.5.1658. PMID 15888843
- [Background] Fass R. Effect of gastroesophageal reflux disease on sleep. J Gastroenterol Hepatol. 2010 May;25 Suppl 1:S41-4. doi: 10.1111/j.1440-1746.2009.06210.x. PMID 20586864
- [Background] Lagergren J, Bergstrom R, Lindgren A, Nyren O. Symptomatic gastroesophageal reflux as a risk factor for esophageal adenocarcinoma. N Engl J Med. 1999 Mar 18;340(11):825-31. doi: 10.1056/NEJM199903183401101. PMID 10080844
- [Background] Elleuch N, Hefaiedh R, Karoui S, Fekih M, Zouiten L, Matri S, Filali A. [Nocturnal gastroesophageal reflux. About a pH metric series]. Tunis Med. 2015 Apr;93(4):223-7. French. PMID 26375738
- [Background] Chey WD, Mody RR, Wu EQ, Chen L, Kothari S, Persson B, Beaulieu N, Lu M. Treatment patterns and symptom control in patients with GERD: US community-based survey. Curr Med Res Opin. 2009 Aug;25(8):1869-78. doi: 10.1185/03007990903035745. PMID 19530980
- [Background] Harvey RF, Gordon PC, Hadley N, Long DE, Gill TR, Macpherson RI, Beats BC, Tottle AJ. Effects of sleeping with the bed-head raised and of ranitidine in patients with severe peptic oesophagitis. Lancet. 1987 Nov 21;2(8569):1200-3. doi: 10.1016/s0140-6736(87)91332-8. PMID 2890820
- [Background] Hamilton JW, Boisen RJ, Yamamoto DT, Wagner JL, Reichelderfer M. Sleeping on a wedge diminishes exposure of the esophagus to refluxed acid. Dig Dis Sci. 1988 May;33(5):518-22. doi: 10.1007/BF01798350. PMID 3359906
- [Background] Johnson LF, DeMeester TR. Evaluation of elevation of the head of the bed, bethanechol, and antacid form tablets on gastroesophageal reflux. Dig Dis Sci. 1981 Aug;26(8):673-80. doi: 10.1007/BF01316854. PMID 7261830
- [Background] Khan BA, Sodhi JS, Zargar SA, Javid G, Yattoo GN, Shah A, Gulzar GM, Khan MA. Effect of bed head elevation during sleep in symptomatic patients of nocturnal gastroesophageal reflux. J Gastroenterol Hepatol. 2012 Jun;27(6):1078-82. doi: 10.1111/j.1440-1746.2011.06968.x. PMID 22098332
- [Background] Stanciu C, Bennett JR. Effects of posture on gastro-oesophageal reflux. Digestion. 1977 Feb;15(2):104-9. doi: 10.1159/000197991. PMID 14044
- [Background] Khoury RM, Camacho-Lobato L, Katz PO, Mohiuddin MA, Castell DO. Influence of spontaneous sleep positions on nighttime recumbent reflux in patients with gastroesophageal reflux disease. Am J Gastroenterol. 1999 Aug;94(8):2069-73. doi: 10.1111/j.1572-0241.1999.01279.x. PMID 10445529
- [Background] Katz LC, Just R, Castell DO. Body position affects recumbent postprandial reflux. J Clin Gastroenterol. 1994 Jun;18(4):280-3. doi: 10.1097/00004836-199406000-00004. PMID 8071510
- [Background] Shay SS, Conwell DL, Mehindru V, Hertz B. The effect of posture on gastroesophageal reflux event frequency and composition during fasting. Am J Gastroenterol. 1996 Jan;91(1):54-60. PMID 8561144
- [Background] van Herwaarden MA, Katzka DA, Smout AJ, Samsom M, Gideon M, Castell DO. Effect of different recumbent positions on postprandial gastroesophageal reflux in normal subjects. Am J Gastroenterol. 2000 Oct;95(10):2731-6. doi: 10.1111/j.1572-0241.2000.03180.x. PMID 11051341
- [Background] Person E, Rife C, Freeman J, Clark A, Castell DO. A Novel Sleep Positioning Device Reduces Gastroesophageal Reflux: A Randomized Controlled Trial. J Clin Gastroenterol. 2015 Sep;49(8):655-9. doi: 10.1097/MCG.0000000000000359. PMID 26053170
- [Background] Allampati S, Lopez R, Thota PN, Ray M, Birgisson S, Gabbard SL. Use of a positional therapy device significantly improves nocturnal gastroesophageal reflux symptoms. Dis Esophagus. 2017 Feb 1;30(3):1-7. doi: 10.1111/dote.12495. PMID 27629558